CLINICAL TRIAL: NCT02216097
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group Phase 2 Study To Assess Effects Of Pf 04457845 On Bold Functional Mri In Subjects With Ptsd
Brief Title: A Study To Assess the Effects Of PF-04457845 On BOLD fMRI In Subjects With Post Traumatic Stress Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study stopped based on Pfizer portfolio prioritization and not due to safety and/or efficacy concern or change in benefit:risk assessment of PF-04457845.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B0541013
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Results first posted 2016-04-08 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-05

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-pyridazin-3-yl-4-(3-((5-(trifluoromethyl)pyridin-2-yl)oxy)benzylidene)piperidine-1-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Drug: PF-04457845
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04457845 — 4mg PF-04457845 tablet taken once daily for 7 days.
  Arms: Treatment
Drug: Placebo — Matching placebo tablet taken once daily for 7 days.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate proof of mechanism of PF-04457845, using a well-established neuroimaging paradigm including behavioral tasks selected to activate neuro-circuitry relevant to Post Traumatic Stress Disorder. It is hypothesized that PF-04457845 will modulate the Blood-oxygen-level dependent Functional Magnetic Resonance Imaging signal from the relevant neuro-circuits in patients with Post Traumatic Stress Disorder.

DETAILED DESCRIPTION:
This is a Phase II, randomized, placebo-controlled, parallel group design study in male and female subjects with moderate-to-severe Post Traumatic Stress Disorder between the ages of 18 and 60 years old. During this study, a dose of 4 mg PF-04457845 will be administered in the morning on Days 1-7. On Each subject will undergo a resting state fMRI (pre and post and day 8), a fearful vs. neutral faces fMRI task and a fear extinction fMRI paradigm. The Emotional Faces Paradigm and resting state tasks will be performed on Day 1 (prior to drug or placebo) and on Day 8. Acquisition of fear conditioning will be performed during the first imaging session on Day 1. After the first imaging session on Day 1, subjects will complete behavioral rating scales and then be dosed. Approximately six hours after dosing subjects will re-enter the scanner and perform the fear extinction paradigm. On Day 2, subjects will perform the fear extinction memory retention task within the scanner. Further physiological monitoring, including skin conductance and heart rate, will take place during the fear extinction paradigm. One safety follow-up visit will occur between Days 11-18.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-60 years of age with a primary psychiatric diagnosis of Post Traumatic Stress Disorder

Exclusion Criteria:

* Other psychiatric illness requiring current treatment with medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Clinical and Translational Science Institute (CTSI), New York, New York
  - NYU CTSI Research Pharmacy (Drug Shipment Address), New York, New York
  - NYU School of Medicine, New York, New York

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0541013&StudyName=A%20Study%20To%20Assess%20Effects%20Of%20PF-04457845%20On%20Blood-Oxygen-Level%20Dependent%20Functional%20Magnetic%20Resonance%20Imaging%20In%20Subjects%20With%20Post%20Traum

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04457845: PF-04457845 4 milligrams (mg) was orally administered once daily in the morning on Days 1 to 7.
- Placebo: Placebo matched to PF-04457845 was orally administered once daily in the morning on Days 1 to 7.
Period: Overall Study
Arm/Group | PF-04457845 | Placebo
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04457845 | Placebo | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.6 (11.4) | 36.2 (15.1) | 35.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Blood-Oxygen-Level Dependent (BOLD) Functional Magnetic Resonance Imaging fMRI) Percent Signal Change in Fearful Versus Neutral Face Contrast in Bilateral Amygdala
Description: Baseline BOLD fMRI percent signal change measured from baseline in fearful versus neutral face contrast during the emotional face processing task in bilateral amygdala.
Time Frame: Baseline, Day 8
Population: There were no efficacy evaluations done in this study because of a change in the planned analysis after the study was prematurely terminated due to Good Clinical Practice (GCP) non-compliance that resulted in data integrity and quality issues.
Arm/Group | PF-04457845 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in BOLD fMRI Percent Activation in Bilateral Ventromedial Pre-Frontal Cortex (vmPFC)
Description: Difference measured in BOLD fMRI percent activation in the bilateral vmPFC during the fear extinction recall phase of the fear extinction paradigm.
Time Frame: Baseline, Day 2
Population: There were no efficacy evaluations done in this study because of a change in the planned analysis after the study was prematurely terminated due to GCP non-compliance that resulted in data integrity and quality issues.
Arm/Group | PF-04457845 | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in BOLD fMRI Percent Signal Change in Fearful Versus Neutral Face Contrast in Right Amygdala
Description: Difference measured in BOLD fMRI percent signal change in the right amygdala in fear versus neutral faces during the emotional face processing task.
Time Frame: Baseline, Day 8
Population: as for outcome 2
Arm/Group | PF-04457845 | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in BOLD fMRI Percent Signal Change in Fearful Versus Neutral Face Contrast in Left Amygdala
Description: Difference measured in BOLD fMRI percent signal change in the left amygdala in fearful versus neutral faces during face processing task.
Time Frame: Baseline, Day 8
Population: as for outcome 2
Arm/Group | PF-04457845 | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: The full physical examination included head, ears, eyes, nose, mouth, skin, heart, and lung examinations, lymph nodes, gastrointestinal, skeletal, and neurological systems.
Time Frame: Baseline to up to Day 18
Population: The safety analysis population included all participants who received study medication.
Measure: Number; unit: participants
Arm/Group | PF-04457845 | Placebo
Number analyzed (Participants) | 8 | 6
participants | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), and Withdrawals Due to AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last study drug administration that were absent before treatment or that worsened relative to pretreatment state. AEs included non-serious AEs and SAEs.
Time Frame: Baseline up to 28 days after last study drug administration (Day 35)
Population: The safety analysis population included all participants who received study medication.
Measure: Number; unit: participants
Arm/Group | PF-04457845 | Placebo
Number analyzed (Participants) | 8 | 6
participants
  Number of Participants with AEs | 6 | 4
  Number of Participants with SAEs | 0 | 0
  Number of Participants Discontinued Due to AEs | 0 | 0

7. Secondary Outcome: Number of Participants With Clinical Laboratory Values Meeting Criteria for Potential Clinical Concern
Description: The following laboratory parameters were analyzed: hematology (hemoglobin, hematocrit, red blood cell count, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes; liver function (aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine, uric acid); electrolytes (sodium, potassium, chloride, calcium, bicarbonate); chemistry (glucose); urinalysis (dipstick) (urine pH, urine glucose, urine protein, urine blood, urine ketones, urine bilirubin, urine nitrite, urine leukocyte esterase); urinalysis microscopy (urine red blood cell, urine white blood cell, urine bacteria). Only parameters with abnormal values were reported.
Time Frame: Baseline up to Day 18
Population: The safety analysis population included all participants who received study medication.
Measure: Number; unit: participants
Arm/Group | PF-04457845 | Placebo
Number analyzed (Participants) | 8 | 6
participants
  Total neutrophils <0.8 times lower limit of normal | 1 | 0
  Urine positive for nitrite | 1 | 0
  Urine positive for leukocyte esterase | 0 | 1

8. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Criteria of Potential Clinical Concern
Description: Vital signs assessment included pulse rate and blood pressure. Criteria for vital sign values meeting potential clinical concern included: supine pulse rate <40 or >120 beats per minute (bpm), standing pulse rate <40 or >140 bpm; systolic blood pressure (SBP) of >=30 millimeters of mercury (mmHg) change from baseline or SBP <90 mmHg; diastolic blood pressure (DBP) >=20 mmHg change from baseline or DBP <50 mmHg.
Time Frame: Baseline up to Day 18
Population: The safety analysis population included all participants who received study medication.
Measure: Number; unit: participants
Arm/Group | PF-04457845 | Placebo
Number analyzed (Participants) | 8 | 6
participants
  Supine SBP <90 mmHg | 0 | 0
  Standing SBP <90 mmHg | 0 | 0
  Supine DBP <50 mmHg | 0 | 0
  Standing DBP <50 mmHg | 0 | 0
  Supine Pulse Rate <40 or >120 bpm | 0 | 0
  Standing Pulse Rate <40 or >140 bpm | 0 | 0
  Supine SBP >=30 mmHg Increase From Baseline | 0 | 0
  Standing SBP >=30 mmHg Increase From Baseline | 0 | 1
  Supine DBP >=20 mmHg Increase From Baseline | 1 | 0
  Standing DBP >=20 mmHg Increase From Baseline | 0 | 0
  Supine SBP >=30 mmHg Decrease From Baseline | 0 | 0
  Standing SBP >=30 mmHg Decrease From Baseline | 0 | 0
  Supine DBP >=20 mmHg Decrease From Baseline | 0 | 0
  Standing DBP >=20 mmHg Decrease From Baseline | 1 | 1

9. Secondary Outcome: Number of Participants With Post-Baseline Electrocardiogram (ECG) Values Meeting Criteria of Potential Clinical Concern
Description: ECG criteria of potential clinical concern were QTc absolute value >=450 milliseconds (msec) or QTc absolute change >=30 msec.
Time Frame: Baseline up to Day 18
Population: The safety analysis population included all participants who received study medication.
Measure: Number; unit: participants
Arm/Group | PF-04457845 | Placebo
Number analyzed (Participants) | 8 | 6
participants
  QTcF Interval 450-<480 msec | 0 | 0
  QTcF Interval 480-<500 msec | 0 | 0
  QTcF Interval >=500 msec | 0 | 0
  QTcF Interval >=30 msec Increase From Baseline | 0 | 0

ADVERSE EVENTS:
Arm/Group | PF-04457845 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 6/8 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-04457845 (N=8) | Placebo (N=6)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 3 (3)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Sleep paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0)
Flashback (Psychiatric disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
There were no efficacy evaluations done in this study because of a change in the planned analysis after the study was prematurely terminated due to GCP non-compliance that resulted in data integrity and quality issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.